CLINICAL TRIAL: NCT04804059
Title: An Open Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-APX001 in Healthy Male Subjects After Oral and Intravenous Dosing
Brief Title: A Study to Assess the Mass Balance Recovery and Metabolite Profile & Identification of [14C]-APX001 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APX001-104; C4791004 (Other: Alias Study Number)
Record Dates: First submitted 2020-10-01; First posted 2021-03-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): [14C]-APX001 Oral Solution
  Interventions: Drug: [14C]-APX001 Oral Solution
- Cohort B (Experimental): [14C]-APX001 Solution for Infusion
  Interventions: Drug: [14C]-APX001 Solution for Infusion

INTERVENTIONS:
Drug: [14C]-APX001 Oral Solution — Total dose containing NMT 3.1 MBq (84.0 µCi) 14C
  Arms: Cohort A
Drug: [14C]-APX001 Solution for Infusion — Total dose containing NMT 3.4 MBq (93.0 µCi) 14C
  Arms: Cohort B

SUMMARY:
This is a single-center, open-label, non-randomized, single dose study in healthy male subjects. It was planned to enroll 2 cohorts of 5 subjects (10 subjects in total), with the target of achieving data in 4 evaluable subjects per cohort. Five subjects were to receive a single oral dose of APX001 and not more than (NMT) 3.1 megabecquerel (MBq) (84.0 microcurie [μCi]) 14C in the fed state. Five subjects were to receive a single IV administration containing APX001 and NMT 3.4 MBq (93.0 μCi) 14C in the fed state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 30 to 65 years of age
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination)
5. Must have been willing and able to communicate and participate in the whole study
6. Must have had regular bowel movements (i.e. average stool production of ≥1 and

   ≤3 stools per day)
7. Must have provided written informed consent
8. Must have adhered to the contraception requirements defined in Section 9.4 of the protocol (Appendix 16.1.1)

Exclusion Criteria:

1. Subjects who had received any IMP in a clinical research study within the previous 3 months or a similar 14C radioactive clinical trial within the previous 12 months
2. Subjects who were study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who had previously been enrolled in this study.
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
6. Current smokers and those who had smoked within the last 12 months. A breath carbon monoxide (CO) reading of greater than 10 ppm at screening and admission
7. Current users of e-cigarettes and nicotine replacement products and those who had used these products within the last 12 months
8. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeded 5 millisieverts (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, was to participate in the study
9. Subjects who did not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator at screening
10. Clinically significant abnormality on electrocardiogram (ECG) as judged by the investigator
11. Clinically significant abnormal biochemistry, hematology or urinalysis at screening as judged by the investigator (laboratory parameters are listed in Appendix 1 of the protocol, Appendix 16.1.1)
12. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1 of the protocol, Appendix 16.1.1)
13. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
14. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
15. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal (GI) disease, neurological or psychiatric disorder, as judged by the investigator
16. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
17. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever was allowed unless it was active
18. Donation or loss of greater than 400 mL of blood within the previous 3 months
19. Subjects who were taking, or had taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration (see Section 11.4 of the protocol, Appendix 16.1.1). Exceptions may have applied on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
20. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery as measured by mass unit equiv/g after a single oral or single intravenous (IV) dose of carbon-14 (14C)-labelled APX001 ([14C]-APX001). | 3 weeks
Profiling of metabolites of [14C]-APX001 in plasma and excreta. | 3 weeks
  Plasma, urine and feces samples from subjects dosed with [14C]-APX001 were analyzed using high resolution, accurate mass liquid chromatography tandem mass spectrometry (LC-MS/MS) with in-line fraction collection and off-line counting to obtain [14C]-radiochromatographic profiles and provide information on the nature of the radioactive components present, including chemical structure identification.

SECONDARY OUTCOMES:
Elimination pathway of [14C]-APX001 following a single oral or single IV dose of [14C]-APX001. | 3 weeks
  Amount of radioactivity recovered from urine and feces over time was measured by liquid scintillation counting (LSC) and expressed as a percentage of administered radioactivity.
Extent of distribution of total radioactivity into blood cells following a single oral or single IV dose of [14C]-APX001. | 3 weeks
  Amount of radioactivity in whole blood over time was quantified by LSC and expressed in ng equivalents free drug/g.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

REFERENCES:
- [Derived] Hodges MR, Ople E, Evans P, Pantophlet AJ(, Richardson J, Williams D, Tripathy S, Tawadrous M, Jakate A. A phase 1 open label study to assess the human mass balance and metabolite profile of 14C-fosmanogepix, a novel Gwt-1 inhibitor in healthy male participants. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0027324. doi: 10.1128/aac.00273-24. Epub 2024 Jul 16. PMID 39012090